CLINICAL TRIAL: NCT01030393
Title: Intra-uterine Injection of Human Chorionic Gonadotrophin Before Embryo Transfer in ICSI
Brief Title: Intra-uterine Injection of Human Chorionic Gonadotrophin (hCG) Before Embryo Transfer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Egyptian IVF-ET Center (Other)
Responsible Party: Principal Investigator, Ragaa Mansour, Director, The Egyptian IVF-ET Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hCG 100
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Infertility
Keywords: hCG; pregnancy; implantation; ICSI; IVF
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intrauterine hCG (Experimental): Experimental arm : intrauterine injection of 100 iu(group1)or 200 iu (group2) of hCG before embryo transfer.
  Intrauterine injection of 500 iu hCG before embryo transfer
  Interventions: Drug: human chorionic gonadotrophin

INTERVENTIONS:
Drug: human chorionic gonadotrophin — intrauterine injection of 100 iu (group1) or 200 iu (group2) of hCG before embryo transfer in IVF/ICSI And intrauterine injection of 500 iu hCG before embryo transfer .
  Other Names: choriomon

SUMMARY:
Chorionic gonadotrophins (hCG) play an important role in implantation. The aim of the study is to evaluate the effect of intrauterine injection of hCG before embryo transfer in IVF/ICSI on the implantation and pregnancy rates. The rational is that intrauterine hCG injection will attract regulatory T cells and improve implantation.

DETAILED DESCRIPTION:
Background :

Human chorionic gonadotrophin ( hCG) was found to secreted immediately after fertilization by the embryo. It plays an important role in implantation and in attracting regulatory T cells to the endometrium.

Rational :

Intrauterine injection of hCG before embryo transfer in IVF/ICSI may increase endometrial regulatory T cells ( Treg ) and improve the implantation and pregnancy rates.

Aim of the work :

To study the effect of intrauterine injection of hCG before embryo transfer on the implantation and pregnancy rates after IVF/ICSI.

Subjects :

Infertile patients undergoing ICSI.

Inclusion criteria :

* Female age less than 40 years
* Male factor infertility
* Normal female hormonal profile and uterine cavity

Exclusion criteria :

* Previous ICSI failure
* Azoospermia
* Endometriosis

Study group: Intrauterine injection of 100 iu of hCG (group 1)or 200 iu of hCG ( group 2) will be done during the dummy embryo transfer which is done 10-15 minutes before the actual embryo transfer.

Control group: The embryo transfer will be done without prior intrauterine injection of hCG

Main outcome measures :

Implantation and pregnancy rates

Secondary outcome measures :

miscarriage and delivery rates

ELIGIBILITY:
Inclusion Criteria:

* male factor infertility
* normal female hormonal profile
* normal uterine cavity

Exclusion Criteria:

* previous ICSI failure
* endometriosis
* azoospermia

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 472 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
implantation and pregnancy rates | 5 weeks after embryo transfer

SECONDARY OUTCOMES:
miscarriage and delivery rates | 9 months from embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ragaa T Mansour, MD,PhD, Principal Investigator — The Egyptian IVF-ET Center
Locations (1):
- The Egyptian IVF- ET center, Cairo, Egypt

REFERENCES:
- [Background] Schumacher A, Brachwitz N, Sohr S, Engeland K, Langwisch S, Dolaptchieva M, Alexander T, Taran A, Malfertheiner SF, Costa SD, Zimmermann G, Nitschke C, Volk HD, Alexander H, Gunzer M, Zenclussen AC. Human chorionic gonadotropin attracts regulatory T cells into the fetal-maternal interface during early human pregnancy. J Immunol. 2009 May 1;182(9):5488-97. doi: 10.4049/jimmunol.0803177. PMID 19380797
- [Derived] Mansour R, Tawab N, Kamal O, El-Faissal Y, Serour A, Aboulghar M, Serour G. Intrauterine injection of human chorionic gonadotropin before embryo transfer significantly improves the implantation and pregnancy rates in in vitro fertilization/intracytoplasmic sperm injection: a prospective randomized study. Fertil Steril. 2011 Dec;96(6):1370-1374.e1. doi: 10.1016/j.fertnstert.2011.09.044. Epub 2011 Nov 1. PMID 22047664